CLINICAL TRIAL: NCT00915031
Title: Hypothermic Nerve Sparing Radical Prostatectomy
Brief Title: Use of Hypothermia During Robotic Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Thomas E. Ahlering, MD, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008-6397
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer
Keywords: Robotic prostatectomy; Hypothermia; Potency
MeSH Terms: conditions — Prostatic Neoplasms; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypothermia Only OR (Active Comparator): Use of Hypothermia Cooling device only in the operating room. Intervention is Hypothermia Cooling Device.
  Interventions: Device: UroCool
- Hypothermia in OR + Recovery (Active Comparator): Use of hypothermia cooling device in the operating room and up to five hours after surgery is intervention.
  Interventions: Device: UroCool

INTERVENTIONS:
Device: UroCool — Hypothermia Endorectal Device

SUMMARY:
Robotic assisted laparoscopic radical prostatectomy (RLP) has gained widespread acceptance as a standard treatment for clinically localized prostate cancer. Despite the enhanced visualization and precise dissection afforded by the robotic platform, two major comorbidities affect a significant number of men: incontinence and erectile function.

Urinary continence and erectile function

It is commonly believed that the most important factor affecting continence is preservation of the external urinary sphincter complex which lies just below the prostate. Trauma to the urethral tissue itself after it is transected from the prostate and damage to the autonomic nerves that control this sphincter may lead to sphincteric dysfunction. In addition, dissection of the bladder may lead to bladder irritability which also plays a role in incontinence. Surgical removal of the prostate also causes significant inflammatory damage to the pelvic floor which likely delays recovery of urinary continence. The same trauma issues apply to sexual function.

One possible method to protect the nerves and other tissues from operative trauma may be the use of local hypothermia (cold-ischemia) to the pelvis. Local tissue hypothermia using ice, ice slush, or cold irrigation has been safely and routinely used for decades in humans during brain, heart, and kidney surgery to minimize organ damage. Yet, this technique has never been applied to prostate surgery. We will accomplish local cooling of the pelvis using a cooling balloon inserted into the rectum. The cooling balloon is powered by an FDA approved cooling system developed by Innercool therapies. Temperatures of 57-86 degrees F (22+/-8 degrees C).

DETAILED DESCRIPTION:
2. 1. Selection of the Patients From June 2002 to August 2015, a total of 1,503 patients underwent RARP. During this period, perioperative data, including postoperative functional outcomes, were prospectively collected using a customized database; our ethics committee approved the data collection. Erectile function was assessed using the sexual health profile for men (SHIM) score at 3, 9, 15, and 24 months and then annually after surgery, and the duration of pad-free continence recovery was asked by a non-physician third party. In our institution, RH was applied during RARP for all patients from February 2008 to March 2015 (consecutively between the 671st and 1459th cases). Among the recruited patients, 789 men (52.6%) underwent HP, leaving the other 711 (47.4%) as controls.

The inclusion criteria for this study were as follows: (1) bilateral nerve-sparing RARP (over 70%) and (2) a minimum follow-up of 15 months. The exclusion criteria were as follows: (1) men with a history of salvage radiation therapy, chemotherapy, or hormone therapy after RARP (n=98) and (2) the presence of a high-risk disease with an initial prostate-specific antigen (PSA) level over 20 ng/ml or biopsy Gleason score over 8, which may influence the refining surgical plane around the neurovascular bundle (NVB), thereby affecting the degrees of nerve-sparing strategy at the time of surgery (n=275). Further, (3) the initial 100 cases were excluded to avoid potential bias from the learning period. From a cohort of 1,503 patients, 59 (3.92%) men whose potency outcome within 15 months was not assessed were also excluded from the study. Finally, 930 patients were selected for the analysis; half of the procedures (n=466, 50.1%) were performed under RH and the remaining other half (n=464, 49.9%) as normothermal controls.

2. 2. Endpoints of the Study The primary endpoints of this study were the SHIM score and the rate of potency regain, which was defined as a SHIM score >17 in the RH and control groups 15 months after surgery. Considering the proven impacts of age and preoperative SHIM scores on the recovery of potency, the groups were further divided into the young and potent (YP: age <65 years and SHIM score ≥22, n=409, 43.9%) subgroup and susceptible for impotency (SI: age ≥65 years or SHIM score <22, n=512, 55.1%) counterpart and investigated the sexual function of the YP subgroup. The secondary endpoints were the duration of pad-free continence regain and the rate of continence recovery within 3 months after surgery, especially in the YP subgroup.

2.3. Surgical Protocol for RH All procedures were performed by a single surgeon. RH was achieved by devising an endorectal cooling balloon system (ECB) as previously reported [2, 4, 5]. In brief, a 40-cm, 24-F, 3-way latex urethral catheter was placed inside a 5 × 2.5-inch elliptic latex balloon that distended at a low pressure and conformed to the rectal wall without excessive deformations. The lubricated ECB was inserted just inside the anus and anchored by inflating the catheter balloon to 20 ml. The ECB was then distended and cycled continuously with cold saline (4°C) by gravity 40 cm above the patient. The ECB volume was ~200 ml. A 9-F esophageal probe (Smiths Medical ASD, Rockland, MA) was used to obtain the intracorporeal temperature readings directly along the anterior surface of the rectum/NVB.

ELIGIBILITY:
Inclusion Criteria:

* adult males
* receiving robotic radical prostatectomy for the treatment of prostate cancer

Exclusion Criteria:

* previous radiation
* previous cryotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Actual)
Dates: Start 2009-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ahlering, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients will be given written and verbal explanation of the study objectives; procedures; potential risks; measures taken to protect confidentiality; any associated costs; alternatives; new findings; and investigator disclosures. Patients will be given time to ask questions.
Groups:
- Hypothermia Only OR: Use of Hypothermia Cooling device only in the operating room
  UroCool: Hypothermia Endorectal Device
- Hypothermia in OR + Recovery: Use of hypothermia cooling device in the operating room and up to five hours after surgery.
  UroCool: Hypothermia Endorectal Device
Period: Overall Study
Arm/Group | Hypothermia Only OR | Hypothermia in OR + Recovery
Started | 714 | 24
Completed | 714 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypothermia Only OR | Hypothermia in OR + Recovery | Total
Number analyzed (Participants) | 714 | 24 | 738
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 246 | 15 | 261
  >=65 years | 468 | 9 | 477
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.677 (7.2) | 62.677 (7.2) | 62.677 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 714 | 24 | 738
Region of Enrollment [Number; unit: participants]
  United States | 714 | 24 | 738

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Safety Using an Improved, More Efficient and Less Labor Intensive Cooling Balloon in Patients Undergoing Hypothermic Nerve-sparing RLP in Participants Determined by Return to Continence
Description: The primary aim is confirmation of the feasibility and safety using an improved, more efficient and less labor intensive cooling balloon in patients undergoing hypothermic nerve-sparing RLP. Continence is defined as no protective urinary pad use as reported by the patient in response to the very first question on page 1 of the sample questionnaire.
Time Frame: During and 6 hours post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hypothermia Only OR | Hypothermia in OR + Recovery
Number analyzed (Participants) | 714 | 24
Participants | 714 | 24

ADVERSE EVENTS:
Time Frame: 5 years
Description: Adverse events were not broken by arm as both groups used the same device and underwent the same procedure leading to a large cohort of patients who underwent cooling. Adverse event reporting was irrespective of arm and cannot be separated. Adverse events were also assessed irrespective of terms.
Groups:
- General Adverse Events: Both arms:
  An adverse event (AE) is any undesirable experience (sign, symptom, significant laboratory abnormality, illness, or other medical event) occurring to a patient that appears or worsens during a clinical study, regardless of etiology.
  * Mild - Awareness of signs or symptoms that are easily tolerated. Signs and symptoms are transient and only of minor irritant type and cause no loss of time from normal activities; symptoms do not require medication or a medical evaluation.
  * Moderate - Discomfort severe enough to cause interference with usual activities. Symptoms may require treatment but not extended hospitalization or intensive care for the patient.
  * Severe - Incapacitating with inability to do work or usual activities. Signs and symptoms may be of systemic nature or require medical evaluation and/or treatment that requires prolonged hospital stay
Arm/Group | General Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/738
Serious Adverse Events (participants affected / at risk) | 0/738
Other Adverse Events (participants affected / at risk) | 2/738
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | General Adverse Events (N=738)
AE1 (Gastrointestinal disorders) | 1 (1) — Disorders involving the gastrointestinal tract, namely the esophagus, stomach, small intestine, large intestine and rectum, and the accessory organs of digestion, the liver, gallbladder, and pancreas.
AE2 (Product Issues) | 1 (1) — Issue with UroCool: Hypothermia Endorectal Device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes